CLINICAL TRIAL: NCT00360672
Title: Phase II Study of Lenalidomide in Patients With Relapsed/Refractory Acute Myelogenous Leukemia or High-Risk Myelodysplastic Syndrome Associated With Chromosome 5 Abnormalities
Brief Title: Revlimid in Patients With Acute Myelogenous Leukemia and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0293
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Revlimid (Experimental): Revlimid 25 mg/day, orally for 21 days with 7 days rest (28 day cycle).
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — 25 mg/day, orally for 21 days with 7 days rest (28 day cycle).
  Other Names: Lenalidomide; CC-5013

SUMMARY:
The goal of this clinical research study is to find out if Revlimid can help to control the disease in patients with relapsed/refractory acute myelogenous leukemia (AML) or high-risk myelodysplastic syndrome (MDS) with abnormalities in chromosome number 5. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Revlimid is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. It is possible that it may help reduce or prevent the growth of cancer cells.

You will have a bone marrow aspiration performed before starting treatment (within 4 weeks) on this study and at about 12 weeks after starting treatment on this study. Your doctor may also decide to perform a bone marrow aspiration before 12 weeks to assess your response to treatment. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

If you are found to be eligible to take part in this study, you will take Revlimid once a day by mouth (with a full glass of water, at least 1 hour before or after a meal) for 21 days.

You will then have 7 days off of the study drug, which is considered a rest period. This entire period is considered 1 cycle of therapy (28 days). The number of treatment cycles you may have will depend on the response of your disease to treatment on this study. You will have blood drawn (about 3 tablespoons) to test for blood counts and chemistries before each treatment cycle. At the end of 3 cycles, your disease will be evaluated for response to the study treatment.

You will be required to return to M. D. Anderson once a month for the first 3 months on this study or as often as the study doctor thinks it is best.

After the first 3 months on this study, you may have blood drawn (about 3 tablespoons) for blood counts and chemistries at your regular doctor's office. The results of your blood tests will then be sent to the research nurse. Your side effects will be reviewed by a doctor or nurse by telephone (in addition to being reviewed in your study diary) before the start of each cycle of treatment. This phone call will last about 10 minutes each time.

You will be taken off this study if your disease gets worse or you experience any intolerable side effects. It is also possible that the study doctor may decide to take you off this study if your disease response is considered less than a complete response. You will have an end-of-study visit, if you are taken off this study for any reason. During the end-of-study visit, you will have blood drawn (about 3 tablespoons) for blood counts and chemistries. You will have an ECG. You may have a urine pregnancy test. You will also have a bone marrow aspiration performed.

This is an investigational study. Revlimid® (lenalidomide) is indicated for the treatment of patients with transfusion-dependent anemia due to Low- or Intermediate-1-risk myelodysplastic syndromes associated with a deletion 5q cytogenetic abnormality with or without additional cytogenetic abnormalities. Revlimid® is also approved in combination with dexamethasone for the treatment of patients with multiple myeloma that have received at least one prior therapy. In this case it will be considered investigational. Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >/= 18 years at the time of signing the informed consent form. (Revlimid has not been tested in younger patients)
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diagnosis of relapsed/refractory AML (other than APL) or high-risk MDS (IPSS categories intermediate-2 and high) with chromosome 5 abnormality as a sole abnormality or with additional abnormalities. MDS patients with blast percentage of >/= 10% will be considered high-risk.
5. All non-hematological toxicity of previous cancer therapy should have resolved to </= grade1 (except alopecia or other toxicities not involving major organs).
6. Should not have received any prior treatment for AML or MDS within 2 weeks of starting Revlimid. Use of hydrea to control proliferative disease will be allowed prior to starting Revlimid and for 7 days during cycles 1 and 2 (Maximum daily dose of 7gm).
7. Eastern Cooperative Oncology Group (ECOG) performance status of </ =2 at study entry
8. Laboratory test results within these ranges: • Serum creatinine </= 1.5 mg/dL • Total bilirubin </=1.5 mg/dL • aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </=2 * upper limit of normal (ULN) or </=5 * ULN if related to disease
9. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International unit (mIU)/mL within 10 - 14 days prior to and again within 24 hours of prescribing Revlimid (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking Revlimid. FCBP must also agree to ongoing pregnancy testing.
10. (continued from above) Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
11. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
12. Disease free of prior malignancies for >/ = 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking Revlimid).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or experimental therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of Revlimid.
8. Concurrent use of other anti-cancer agents or treatments. (Use of hydrea permitted as indicated in inclusion criterion 6)
9. Known positive for HIV or infectious hepatitis type B or C.
10. Heart rate less than or equal to 50.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 08/03/2006 through 05/10/2012. All participants recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Revlimid
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Revlimid
Number analyzed (Participants) | 27
Age Continuous [Median (Full Range); unit: years] | 64 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response (Complete Remissions (CR), Complete Remissions With Incomplete Platelet Recovery [CRp] and Partial Responses)
Description: Response for Acute Myeloid Leukemia (AML) according to 2003 International Working Group (IWG) criteria: CR required absolute neutrophil count (ANC) >1 * 10^9/L, platelet count ≥100 * 10^9/L, < 5% of blast cells in bone marrow. CRp: as above except platelet count <100 * 10^9/L. Partial remission: as CR except for presence of 5-25% marrow blasts and with a decrease of marrow blast at least 50%. Response for Myelodysplastic Syndrome (MDS) was defined based on the 2006 IWG criteria. All participants with MDS who achieved hematological CR, Partial Response (PR), marrow CR, and hematological improvement considered responders.
Time Frame: Following three 28-day cycles evaluated for response
Measure: Number; unit: participants
Arm/Group | Revlimid
Number analyzed (Participants) | 27
participants
  Complete Remission | 1
  Complete Remission Incomplete Platelet Recovery | 1
  Partial Remission | 0

ADVERSE EVENTS:
Time Frame: 5 years, 8 months
Arm/Group | Revlimid
Serious Adverse Events (participants affected / at risk) | 9/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid (N=27)
Infection (Infections and infestations) | 3 (3)
Vomit (Gastrointestinal disorders) | 1 (1)
Hemorrhage (Gastrointestinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (3)
Death (General disorders) | 5 (5)
Renal Failure (Renal and urinary disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid (N=27)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (14)
Neutropenic Fever (Infections and infestations) | 4 (4)
Neutropenic Fever With Pneumonia (Infections and infestations) | 3 (3)
Nonneutropenic Infection (Infections and infestations) | 13 (13)
Fatigue (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes